CLINICAL TRIAL: NCT05636631
Title: The Role of Chest Ultrasound in Differentiating Lung Congestion and Pneumonia in Adult Critically-ill Patients and Its Prognostic Impact
Brief Title: Chest U/S in Differentiating Lung Congestion & Pneumonia in Adult Critically-ill Patients and Its Prognostic Impact
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nardin Aymn Boshra, Doctor, Assiut University
Other Study IDs: chest US for lung conditions
Record Dates: First submitted 2022-11-04; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Pneumonia; Pulmonary Edema
MeSH Terms: conditions — Pneumonia; Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Pneumonia (1): Patients presented with symptoms suggestive of pneumonia as fever, tachypnea, cough with sputum. These patients will receive IV fluids & antibiotics with follow up of sepsis parameters
  Interventions: Device: Chest ultrasound
- Patients with decongestive heart failure (2): Patients presented with symptoms suggestive of acute congestive heart failure as dyspnea, orthopnea, bilateral lower limb edema. These patients will receive anti-failure treatment as diuretics, ACE inhibitors & Beta blockers with follow up of resolving signs of decompensated heart failure
  Interventions: Device: Chest ultrasound

INTERVENTIONS:
Device: Chest ultrasound — chest ultrasound as a non invasive, low cost & bedside device for differentiation & follow up of lung congestion & pneumonia

SUMMARY:
This study aim will be to assess the effectiveness of chest ultrasound as a diagnostic and differentiating modality in cases of pneumonia and lung congestion . It also evaluates chests sonography effectiveness in follow-up of patients with pneumonia and lung congestion .

DETAILED DESCRIPTION:
Lung ultrasound (LUS) is used at the bedside in emergency and critical care settings. It is a rapid and low-cost approach that can direct patient care without the use of harmful radiation. The success of this technique depends on its simplicity to discover the sonographic signs which indicate certain lung pathology. These signs include a hyperechoic and sliding line, moving forward and back with ventilation seen 0.5 cm below the rib line and is called the pleural line. The A-profile associates anterior lung sliding with A lines. A lines are horizontal repetition artifacts of the pleural line. The B-profile associates anterior lung sliding with B lines. B lines appear as shining vertical lines arising from the pleural line and reach the edge of the screen.

Several pathological etiologies can fill the alveolar spaces, with fluid (heart failure), pus (pneumonia which is the commonest), blood (pulmonary hemorrhage), and cells (lung cancer).

Other causes of lung consolidation may include atelectasis, pulmonary edema, infarction, and lung cancer. Chest imaging with CT is regarded as the gold standard modality allowing for the diagnosis of pneumonia in earlier stage and with higher sensitivity and specificity. On the contrary, cardiogenic pulmonary edema (CPE) is defined as alveolar transudation caused by elevated pulmonary capillary hydrostatic pressure secondary to increased pulmonary venous pressure with low-protein content in the interstitial tissue of lung as a result of cardiac dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Adult (above 18 years old)
* Both genders
* Patient with symptoms suggestive of pneumonia
* Patient with symptoms suggestive of acute congestive heart failure
* admitted to Critical care unit

Exclusion Criteria:

* Patients with Renal induced lung congestion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: both genders adult (above age of 18 years) critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic tool | Baseline
  Diagnosis of pneumonia vs lung congestion by using chest ultrasound examination viewing A-lines, B-lines, pleural effusion presence & its initial amount .
Follow up after initiation of treatment | Baseline ( day 3 of hospital admission)
  Follow up of findings of chest U.S on day 1 after initiating therapy using same parameters ( A-lines, B-lines, pleural effusion) on day 3 of hospital admission
Follow up before assessing final outcome | Baseline ( day 7 of hospital admission)
  Follow up of findings of chest U.S on day 1 after initiating therapy using same parameters ( A-lines, B-lines, pleural effusion) on day 7 of hospital admission

SECONDARY OUTCOMES:
morbidity & mortality | baseline
  if patient's symptoms improved or not If patient died or not

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ashry, Professor, Study Director — Professor Faculty of Medicine, Assiut University
Locations (1):
- Nardin Aymn, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Volpicelli G, Cardinale L, Garofalo G, Veltri A. Usefulness of lung ultrasound in the bedside distinction between pulmonary edema and exacerbation of COPD. Emerg Radiol. 2008 May;15(3):145-51. doi: 10.1007/s10140-008-0701-x. Epub 2008 Jan 31. PMID 18236088
- [Background] Lichtenstein DA. BLUE-protocol and FALLS-protocol: two applications of lung ultrasound in the critically ill. Chest. 2015 Jun;147(6):1659-1670. doi: 10.1378/chest.14-1313. PMID 26033127